CLINICAL TRIAL: NCT00431574
Title: Antipsychotic Medication Extended Dosing Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 234/2003
Record Dates: First submitted 2007-02-02; First posted 2007-02-06 (Estimated); Last update posted 2024-02-07 (Actual); Status verified 2008-02

CONDITIONS: Schizophrenia
Keywords: schizophrenia; schizoaffective; antipsychotic; randomized control trial
MeSH Terms: conditions — Schizophrenia | interventions — Biomarkers, Pharmacological

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

INTERVENTIONS:
Procedure: dosing

SUMMARY:
In patients stabilized on their antipsychotic and demonstrating evidence of good clinical response, there will not be a significant change in symptoms if their medication is decreased to every 2 days rather than daily. This decrease in antipsychotic exposure will lead to a reduction in side effects, as well as improved subjective response to treatment.

DETAILED DESCRIPTION:
The present study is a 6-month, double-blind study of patients with schizophrenia stabilized on their current antipsychotic (monotherapy) for a period of at least 3 months. After providing informed consent, individuals will be randomly assigned to 1 of 2 treatment arms: regular daily antipsychotic dosing or active medication at the same daily dose every 2nd day. Various scales to measure clinical response and side effects will be administered at baseline, as well as every 2 weeks thereafter. Subjective scales will also be employed, and lab evaluations will include plasma antipsychotic levels at baseline and endpoint, as well as prolactin. Our sample size will be 20/group.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of schizophrenia or schizo-affective disorder
* Capacity to provide written, informed consent
* Stabilized* on a single oral antipsychotic for at least three months (excluding CLOZAPINE or QUETIAPINE)
* Evidence of compliance with previous antipsychotic treatment, i.e. greater than 90% * defined as 2 consecutively identical CGI evaluations (screening and baseline, at least one week apart)

Exclusion Criteria:

* exposure to depot antipsychotic during 12 months prior to enrollment
* substance-related disorders according to DSM-IV

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2002-08; Primary Completion 2007-06 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Clinical Global Impression every 2 weeks
Simpson and Angus Rating Scale for Extrapyramidal Effects every 2 weeks
Barnes Rating Scale for Drug-Induced Akathisia every 2 weeks
Abnormal Involuntary Movement Scale every 2 weeks
Drug Attitude Inventory every 2 weeks
Calgary Depression Scale for Schizophrenia every 2 weeks
Brief Psychiatric Rating Scale every 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gary J Remington, MD, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Remington G, Seeman P, Feingold A, Mann S, Shammi C, Kapur S. "Extended" antipsychotic dosing in the maintenance treatment of schizophrenia: a double-blind, placebo-controlled trial. J Clin Psychiatry. 2011 Aug;72(8):1042-8. doi: 10.4088/JCP.09m05866yel. Epub 2010 Sep 7. PMID 20868639